CLINICAL TRIAL: NCT06046079
Title: A Mixed Methods Study of the Association Between LAI PrEP Initiation and Adherence, and Utilization of Health and Social Support Services Among Key Populations in Washington DC
Brief Title: Predictors of Health Service Utilizations Among Key Population in Washington DC
Status: Recruiting | Type: Observational
Sponsor: Us Helping Us, People Into Living, Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: HOPP1
Record Dates: First submitted 2023-09-13; First posted 2023-09-21 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Pre-exposure Prophylaxis; HIV; Health Behavior
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The primary objective of the proposed study is to investigate how PrEP use might result in an increase in the utilization of health and social services offered at a local community-based organization. Our primary hypothesis is that the investigators will observe higher utilization of sexual health (STI screenings), psychosocial health (psychotherapy, and substance use treatment) and other social services (emergency cash assistance, food pantry, transportation assistance, clothing,and housing resources) among PrEP users (LAI-PrEP or daily oral) compared to participants who are PrEP naïve over the 12-month follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* age of 18 years or above;
* confirmed HIV-negative status;
* residence in the Washington, DC metropolitan area;
* one of the following PrEP profiles (PrEP naïve [no history of any PrEP use in the past] currently on daily oral PrEP or receiving LAI-PrEP).

Exclusion Criteria:

* being younger than18 years of age
* being unable to speak and/or read English
* a reported residence outside of the defined Washington, DC metropolitan area
* being unable or unwilling to provide written informed consent
* being unable to comply with the requirements of the protocol (i.e. persons with mental health conditions, persons who are intoxicated or incoherent for other reasons)
* evidence of suspected hepatoxicity

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Black sexual minority men, Latino sexual minority men, Black cisgender women, people who inject drugs, and transgender women
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-08-25 (Actual); Primary Completion 2025-07-03 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
The rate of service utilization (sexual health, psychosocial health & other social services) over 12 months as a function of demographic characteristics, mental health, and substance use behavior. | Over 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Us Helping Us, People into Living Inc, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: Undecided